CLINICAL TRIAL: NCT03784417
Title: EUS-guided Laser Complete Ablation of Advanced Pancreatic Ductal Adenocarcinoma: a Feasibility Study
Brief Title: EUS-guided Laser Ablation in Pancreatic Adenocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: device unavalaible
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUS-LASER
Record Dates: First submitted 2018-11-25; First posted 2018-12-21 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Adenocarcinoma; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-guided laser ablation (Experimental): Laser ablation will be performed using a 1064-nm wavelength laser with the insertion of a 300-μm optical fiber through a 22-gauge needle under endoscopic ultrasonography guidance.
  Interventions: Device: EUS-guided laser ablation

INTERVENTIONS:
Device: EUS-guided laser ablation — EUS-guided LA will be performed with an endoscopic ultrasound guided approach using a 1064-nm wavelength laser with the insertion of a 300-μm optical fiber through a 22-gauge flexible needle that is inserted in the working channel of the echoendoscope.

SUMMARY:
This study evaluates the possibility of performing local therapy for PDAC using laser ablation of the tumor under ultrasonography (EUS) guidance.

Safety of the procedure as well as post procedural quality of life will be also evaluated.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) is projected to be the second cause of cancer death in Western societies within a decade. Management include chemotherapy and/or radiation therapy, while resectable disease is possible only in 15% of cases.

Despite these therapeutic approaches, the survival rate of unresectable pancreatic cancer remains disappointing. Recently, there is a growing interest in the development of alternative therapeutic approaches, which can work in parallel with standard chemoradiation therapy. These methods include intra-lesion injection/instillation of antitumoral agents performed through a laparoscopic approach, or percutaneously or under endoscopic ultrasound (EUS) guidance and tumor volume reduction procedures using ablative techniques.

In this context laser ablation has been reported to be effective in inducing coagulative necrosis of the tumour in absence of major adverse events. However, the available studies on the matter are limited by small sample size, lack of extended follow up and informations about the possibility to ablate the entire tumour mass.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of pancreatic ductal adenocarcinoma
* Unresectable advanced, non-metastatic Stage III tumor
* Stable disease without regression or progression after 6 months of chemotherapeutic treatment
* Locally progressive disease after chemiotherapy, without evidence of metastases
* Age >18 and <80 years
* Willing to be followed up c/o the Fondazione Policlinico A. Gemelli University Hospital
* Signed informed consent

Exclusion Criteria:

* Stage I, Stage II, Stage IV disease
* Absolute contraindications to general anesthesia or deep sedation
* Absolute contraindications to perform digestive endoscopy
* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma (FFP)
* Use of anticoagulants that cannot be discontinued
* International Normalized Ratio (INR) >1.5 or platelet count <50.000
* Pregnancy or lactation
* Unable to sigh informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Tumor necrosis induction by EUS-guided laser ablation (LA) - Number of patients with necrosis of the tumor | at 1 month from the intervention
  Number of patients with necrosis of the tumor, as demonstrated by the involution of the pancreatic mass on CT scan performed after one month from the treatment

SECONDARY OUTCOMES:
Incidence of early and late adverse events after EUS-guided laser ablation (LA) | at 7 days and 3 months from the intervention
  Percentage of early and late adverse events. Early adverse events will be those occurring during the procedure up to the first week after the ablation treatment. Late adverse events will be defined as any adverse event potentially related to the procedure occurring at the site of the primary tumor within 3 months after EUS LA treatment. Adverse events will be considered major if they prevent completion of the scheduled procedure and/or resulted in prolongation of hospital stay, another therapeutic procedure (needing sedation/anesthesia), or subsequent medical consultation. Any potential adverse event such as pancreatitis, burns of the gastric or duodenal walls, bowel injury, or peritonitis will be recorded and graded according to the above-mentioned classification.
Disease response to EUS-guided laser ablation (LA) | From date of treatment, every 4 months, assessed until death or up to 2 years
  Correlation between RNA markers evaluated by TaqMan RNA assay in serum and treatment response
Post-procedural quality of life | From date of enrollment (baseline), every 2 months, assessed until death or up to 2 years
  Change from baseline in quality of life (QOL) scores after treatment evaluated by using the European Organization for Research and Treatment core quality of life questionnaire (EORTC QLQ-C30), version 3.0. EORTC QLQ-C30 questionnaire evaluates 5 functions physical,role,cognitive, emotional, and social), 9 symptoms (fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties) and the global health status. Questions regarding functions and symptoms are scored 1 to 4, with higher values representing a worse outcomes. Questions regarding global health status are scored 1 to 7, with higher values representing better outcomes.
Progression-free-survival (PFS) | From date of enrollment assessed until death or up to 2 years
  PFS defined as the time from the date of trial entry until disease progression or relapse.
Overall survival | From date of enrollment assessed until death or up to 2 years
  Overall survival defined as the length of time (in days) between the treatment date and the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM
  - Universita' Cattolica del Sacro Cuore, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon-Dseagu VL, Devesa SS, Goggins M, Stolzenberg-Solomon R. Pancreatic cancer incidence trends: evidence from the Surveillance, Epidemiology and End Results (SEER) population-based data. Int J Epidemiol. 2018 Apr 1;47(2):427-439. doi: 10.1093/ije/dyx232. PMID 29149259
- [Background] Ryan DP, Hong TS, Bardeesy N. Pancreatic adenocarcinoma. N Engl J Med. 2014 Nov 27;371(22):2140-1. doi: 10.1056/NEJMc1412266. No abstract available. PMID 25427123
- [Background] Lakhtakia S, Seo DW. Endoscopic ultrasonography-guided tumor ablation. Dig Endosc. 2017 May;29(4):486-494. doi: 10.1111/den.12833. Epub 2017 Mar 16. PMID 28171697
- [Background] Han J, Chang KJ. Endoscopic Ultrasound-Guided Direct Intervention for Solid Pancreatic Tumors. Clin Endosc. 2017 Mar;50(2):126-137. doi: 10.5946/ce.2017.034. Epub 2017 Mar 30. PMID 28391669
- [Background] Girelli R, Frigerio I, Salvia R, Barbi E, Tinazzi Martini P, Bassi C. Feasibility and safety of radiofrequency ablation for locally advanced pancreatic cancer. Br J Surg. 2010 Feb;97(2):220-5. doi: 10.1002/bjs.6800. PMID 20069610
- [Background] Girelli R, Frigerio I, Giardino A, Regi P, Gobbo S, Malleo G, Salvia R, Bassi C. Results of 100 pancreatic radiofrequency ablations in the context of a multimodal strategy for stage III ductal adenocarcinoma. Langenbecks Arch Surg. 2013 Jan;398(1):63-9. doi: 10.1007/s00423-012-1011-z. Epub 2012 Sep 29. PMID 23053459
- [Background] Kim HJ, Seo DW, Hassanuddin A, Kim SH, Chae HJ, Jang JW, Park DH, Lee SS, Lee SK, Kim MH. EUS-guided radiofrequency ablation of the porcine pancreas. Gastrointest Endosc. 2012 Nov;76(5):1039-43. doi: 10.1016/j.gie.2012.07.015. PMID 23078928
- [Background] Francica G, Petrolati A, Di Stasio E, Pacella S, Stasi R, Pacella CM. Effectiveness, safety, and local progression after percutaneous laser ablation for hepatocellular carcinoma nodules up to 4 cm are not affected by tumor location. AJR Am J Roentgenol. 2012 Dec;199(6):1393-401. doi: 10.2214/AJR.11.7850. PMID 23169736
- [Background] Di Matteo F, Martino M, Rea R, Pandolfi M, Rabitti C, Masselli GM, Silvestri S, Pacella CM, Papini E, Panzera F, Valeri S, Coppola R, Costamagna G. EUS-guided Nd:YAG laser ablation of normal pancreatic tissue: a pilot study in a pig model. Gastrointest Endosc. 2010 Aug;72(2):358-63. doi: 10.1016/j.gie.2010.02.027. Epub 2010 Jun 11. PMID 20541187
- [Background] Carrara S, Arcidiacono PG, Albarello L, Addis A, Enderle MD, Boemo C, Campagnol M, Ambrosi A, Doglioni C, Testoni PA. Endoscopic ultrasound-guided application of a new hybrid cryotherm probe in porcine pancreas: a preliminary study. Endoscopy. 2008 Apr;40(4):321-6. doi: 10.1055/s-2007-995595. PMID 18389449
- [Background] Di Matteo FM, Saccomandi P, Martino M, Pandolfi M, Pizzicannella M, Balassone V, Schena E, Pacella CM, Silvestri S, Costamagna G. Feasibility of EUS-guided Nd:YAG laser ablation of unresectable pancreatic adenocarcinoma. Gastrointest Endosc. 2018 Jul;88(1):168-174.e1. doi: 10.1016/j.gie.2018.02.007. Epub 2018 Feb 13. PMID 29452076
- [Background] Di Matteo F, Picconi F, Martino M, Pandolfi M, Pacella CM, Schena E, Costamagna G. Endoscopic ultrasound-guided Nd:YAG laser ablation of recurrent pancreatic neuroendocrine tumor: a promising revolution? Endoscopy. 2014;46 Suppl 1 UCTN:E380-1. doi: 10.1055/s-0034-1377376. Epub 2014 Sep 25. No abstract available. PMID 25254586
- [Background] Gress TM, Lausser L, Schirra LR, Ortmuller L, Diels R, Kong B, Michalski CW, Hackert T, Strobel O, Giese NA, Schenk M, Lawlor RT, Scarpa A, Kestler HA, Buchholz M. Combined microRNA and mRNA microfluidic TaqMan array cards for the diagnosis of malignancy of multiple types of pancreatico-biliary tumors in fine-needle aspiration material. Oncotarget. 2017 Nov 21;8(64):108223-108237. doi: 10.18632/oncotarget.22601. eCollection 2017 Dec 8. PMID 29296236
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390